CLINICAL TRIAL: NCT06823700
Title: A Prospective, Multicenter, Single Arm Study to Evaluate the Safety and Effectiveness of Shenqi Transcatheter Mitral Valve Clips Delivery System and Steerable Guide Catheters in Patients with Functional Mitral Regurgitation
Brief Title: Safety and Effectiveness Study of SQ-Kyrin System for Functional Mitral Regurgitation in EU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Shenqi Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVRP01-001C
Record Dates: First submitted 2024-05-30; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Functional Mitral Regurgitation

STUDY DESIGN:
Intervention Model Description: Device: SQ-Kyrin Transcatheter Mitral Valve Repair System
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SQ-Kyrin TMVr System (Experimental)
  Interventions: Device: SQ-Kyrin Transcatheter Mitral Valve Repair System

INTERVENTIONS:
Device: SQ-Kyrin Transcatheter Mitral Valve Repair System — To percutaneously repair the mitral valve via the femoral vein and atrial septum, offering a treatment for symptomatic functional mitral regurgitation through edge-to-edge valve clipping.

SUMMARY:
The investigation objective of this study is to evaluate the safety and effectiveness of the Transcatheter Mitral Valve Clip Delivery System and Steerable Guide Catheter in the population of FMR patients and the accessories devices when used in conjunction with the Transcatheter Mitral Valve Clip Delivery System and Steerable Guide Catheter.

DETAILED DESCRIPTION:
The primary objective is to verify the safety and effectiveness of the Transcatheter Mitral Valve Clip Delivery System and Steerable Guide Catheter produced by Shanghai Shenqi Medical Technology Co., Ltd. In the treatment of patients with moderate-severe (3 +) or severe (4 +) FMR whose symptoms and MR severity persist despite maximally tolerated GDMT as determined by a multidisciplinary heart team experienced in the evaluation and treatment of heart failure and mitral valve disease.

ELIGIBILITY:
Inclusion Criteria:

1. Participant who has provided written informed consent for the investigation.
2. Age ≥18 years.
3. Patients diagnosed with FMR.
4. MR severity is (functional) ≥3+ as determined by transthoracic echocardiography (TTE).
5. LVEF ≥20% to ≤60%.
6. Symptom status: NYHA functional class II to IV despite a stable maximally tolerated GDMT regimen as per guidelines.
7. According to the judgment of local cardiology team, subjects have undergone adequate treatment for at least 30 days (preferably 90 days) based on the criteria recommended in the heart failure guidelines.
8. Subject fulfils FMR anatomy selection criteria.
9. According to the judgment of the local Cardiovascular medical-surgery team, subjects who have high or prohibitive risk for open heart surgery.
10. Left ventricular end-systolic diameter (LVESD)≤70mm.
11. The MR beam mainly originates from the A2/P2 area.
12. Mitral valve coaptation depth≤11mm, coaptation height≥2mm, effective length of anterior and posterior leaflets>10mm.
13. Mitral valve effective orifice area (EOA) ≥ 4.0cm2.
14. No obvious calcification of main grasp mitral valve leaflets.
15. Patient anatomy allows atrial septum approach.

Exclusion Criteria:

1. Life expectancy <1 year due to non-cardiac conditions or heart failure deemed suitable for palliative treatment.
2. Hypotension (systolic pressure <90 mm Hg) or requirement for inotropic support or mechanical hemodynamic support.
3. UNOS status 1 heart transplantation or prior orthotopic heart transplantation.
4. Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology.
5. Fixed pulmonary artery systolic pressure >70 mm Hg.
6. Physical evidence of right-sided congestive heart failure with echocardiographic evidence of moderate or severe right ventricular dysfunction.
7. Mitral valve anatomy which may preclude proper device treatment.
8. Mitral valve area < 4.0 cm2 (if new device therapy may further decrease the mitral orifice area).
9. Any prior mitral valve surgery or transcatheter mitral valve procedure.
10. Stroke or transient ischemic event within 30 days before enrolment.
11. Modified Rankin ≥ Scale 4 disability.
12. Severe symptomatic carotid stenosis (>70% by ultrasound).
13. Need for emergent or urgent intervention for any reason or any planned cardiac intervention within the next 12 months.
14. Implant or revision of any rhythm management device (CRT or CRT-D) or implantable cardioverter-defibrillator within 1 month before enrolment.
15. Untreated clinically significant coronary artery disease requiring revascularization.
16. Any percutaneous cardiovascular intervention, cardiovascular intervention, or carotid intervention within 30 days
17. Tricuspid valve disease requiring intervention or severe or more tricuspid regurgitation.
18. Aortic valve disease requiring intervention or any concomitant treatment.
19. Need for any cardiovascular intervention (other than for MV disease).
20. Echocardiographic evidence of intracardiac mass, thrombus, or vegetation.
21. Active endocarditis.
22. Active infections requiring current antibiotic therapy.
23. Subjects in whom transoesophageal echocardiography is contraindicated or high risk.
24. Any condition making it unlikely the patient will be able to complete all protocol procedures (including compliance with guideline directed medical therapy) and follow-up visits.
25. Patient unable or unwilling to provide written, informed consent before study enrolment.
26. Pregnant woman or woman planning to become pregnant.
27. Patients with severe liver, renal or pulmonary disease, which in investigator opinion may have an impact on patient safety.
28. Clinically significant lab abnormalities which in investigator opinion may have an impact on patient safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with composite measures- All-cause death and recurrent hospitalizations due to heart failure | 12 months
  A composite of all-cause death and recurrent hospitalizations due to heart failure

SECONDARY OUTCOMES:
Technical success rate | immediately after intervention
  Defined by the following four conditions:
  1. No procedural mortality. 2. Successful delivery, implant, retrieval of the delivery system. 3. Successful devices release. 4. No need for any emergency surgery related to the device or surgical approach.
Device success rate | 30 days
  Defined by the following three conditions:
  1. Technical success maintained at day 30. 2. Transthoracic echocardiographic assessment showing MR ≤2+ without significant mitral stenosis. 3. No structural or functional failure of the device.
Procedural success rate | 30 days
  Defined by following two conditions:
  1. Device success. 2. No major adverse events occurred.
The rate of New York Heart Association (NYHA) heart function class I or II | On the day of discharge, 30 days, 6 months, and 12 months
Improvement in quality of life from baseline | 12 months
  Improvement in quality of life (QoL) at 12 months over baseline, as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) score, scale from 0 - 100, and higher scores mean a better outcome.
Rate of MR 2+ or less than 2+ | 30 days, 6 months, and 12 months
  Mitral regurgitation severity grade 2+ or less than 2+
Change from baseline to discharge in MR severity assessed by echocardiography. | On the day of discharge
Rate of hospitalization for heart failure | 30 days, 6 months, and 12 months
Improvement by ≥ 50m in 6-minute walk distance from baseline | 12 months
Improvement in left ventricular end-diastolic volume (LVEDV) from baseline | 12 months
Incidence of all-cause mortality | 30 days, 6 months, and 12 months
Cardiovascular-related mortality | 30 days, 6 months, and 12 months
Incidence of major adverse events | 30 days and 12 months
  The major adverse event refers to the composite endpoint of death, stroke, myocardial infarction, and cardiovascular surgery due to device- or interventional-related adverse events that occurred since successful transfemoral vein puncture and establishment of atrial septal pathway.

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio J Amat-Santos, MD, Ph.D, Principal Investigator — Hospital Clínico Universitario de Valladolid
Locations (1):
- Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No